CLINICAL TRIAL: NCT04170933
Title: A Prospective Study: Magnetic Compression Anastomosis for Recanalization of Biliary Stricture
Brief Title: Magnetic Compression Anastomosis for Recanalization of Biliary Stricture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF-CRF-2015-001-4
Record Dates: First submitted 2019-11-15; First posted 2019-11-20 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-04

CONDITIONS: Biliary Anastomotic Stricture; Biliary Tract Diseases; Cholestasis, Extrahepatic; Endotoxicosis
Keywords: Magnetic recanalization; Biliary Anastomotic Stricture; Biliary Tract Diseases; Cholestasis, Extrahepatic
MeSH Terms: conditions — Biliary Tract Diseases; Cholestasis, Extrahepatic

STUDY DESIGN:
Intervention Model Description: A prospective study of magnetic recanalization in treatment of biliary stricture
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magnetic recanalization (Experimental): The subjects in this group will be treated by magnetic recanalization
  Interventions: Procedure: Magnetic recanalization

INTERVENTIONS:
Procedure: Magnetic recanalization — 1. Establish a percutaneous transhepatic cholangio drainage (PTCD) fistula.
  2. Perform endoscopic sphincterotomy (EST).
  3. Place one magnet above the stricture through the PTCD fistula.
  4. Introduce another magnet below the stricture through the common bile duct with ERCP.
  5. Place the magnets at the appropriate point to attract each other.
  6. The patient will be strictly followed, and the magnets will be taken out out of the mouth by the thread connected with the magnets.
  7. A plastic stent will be placed in the bile duct for lasting support.

SUMMARY:
Biliary stricture is a common complication after end-to-end biliary anastomosis, especially after liver transplantation. This study is designed to investigate the safety and efficacy of magnetic recanalization technique, a newly clinical method, for treating biliary anastomotic stricture.

DETAILED DESCRIPTION:
Biliary anastomotic stricture is a common complication of after end-to-end biliary anastomosis. Magnetic recanalization is a promising way to establish connection of biliary tract after stenosis or completed obstruction. This study is designed to investigate the safety and efficacy of magnetic recanalization among patients with severe biliary stricture after biliary anastmosis. Patients who failed to undergo stent placement with endoscopic retrograde cholangiopancretography (ERCP) would be enrolled for magnetic recanalization treatment. Magnetic treatment will be implemented by several steps. Firstly, placement of one magnet through the sinus of percutaneous transhepatic cholangio drainage (PTCD) in upper part of the bile duct; Second, introduction of another magnet via ERCP into the distal part of the bile duct, and making them be mated together; Third, after necrosis of the tissue between the two magnets, the magnets will drop off and be taken out together through the thread connected with them out of the mouth. Last, a plastic stent should be placed in the bile duct for a lasting support. The time of recanalization (drop off of the magnets), and adverse events (e.g. fever, melena, nausea, vomiting, anorexia, hematemesis, abdominal pain, and gastrointestinal bleeding) will be recorded, and each patient will be followed up for long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years old and ≤65 years old
* 2. patients with biliary stricture after end-to-end biliary anastomosis

Exclusion Criteria:

* 1. Pregnant woman
* 2.Have a history of cardiovascular disease, including coronary heart disease (angina pectoris, myocardial infarction, coronary angiogenesis or electrocardiographic abnormal Q wave (ECG)), stroke (ischemic or hemorrhagic, including transient ischemic attack)
* 3. Severe lung diseases such as COPD and asthma
* 4. Patients with acute infection or inflammation (i.e. pneumonia)
* 5. Any other medical condition considers the longest survival time to be less than 2 years
* 7. Immunodeficiency or HIV positive
* 8. No autonomy, inability to participate in follow-up
* 9. Illiterate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Time duration of biliary recanalization, d (days) | From date of treatment (two magnets mated together) until the date of drop-off or the two magnets from the biliary tract or date of death from any cause, whichever came first, assessed up to 12 months
  Time period for recanalization of the bile duct

SECONDARY OUTCOMES:
Incidence of stricture recurrence | From date of drop-off of the two magnets until the date of biliary stricture recurrence or end of the follow-up or date of death from any cause, whichever came first, assessed up to 12 months
  Incidence of biliary stricture recurrence after magnetic recanalization treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yi Lv, MD,phD, Principal Investigator — First Affiliated Hospital of Xian JiaotongUniversity
Locations (1):
- First Affiliated Hospital of Xian JiaotongUniversity, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided